CLINICAL TRIAL: NCT00340691
Title: Treatment of Mansonella Perstans Infection in an Area Coendemic for Lymphatic Filariasis: A Pilot Study of the Effects of Doxycycline
Brief Title: Doxycycline to Treat Mansonella Perstans Infection in Patients With and Without Lymphatic Filariasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Amy Klion, M.D./National Institute of Allergy and Infectious Diseases, National Institutes of Health
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 999905053; 05-I-N053
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2008-11-25

CONDITIONS: Mansonella Perstans Infection; Mp Microfilaremia
Keywords: Parasite; Chemotherapy; Wuchereria Bancrofti
MeSH Terms: conditions — Mansonelliasis | interventions — Doxycycline

INTERVENTIONS:
Drug: Doxycycline

SUMMARY:
This study will examine: 1) the safety and effectiveness of the drug doxycycline in reducing the number of Mansonella perstans (Mp) worms in the blood of infected patients, and 2) the effects of doxycycline followed by albendazole and ivermectin treatment for lymphatic filariasis, caused by the parasitic worm Wuchereria bancofti (Wb).

Both Mp and Wb very small filarial worms that are spread by mosquitoes. Some people are infected with both Mp and Wb. Although most people do not become ill from infection with these parasites, some develop symptoms. Wb can cause swellings in the arms, legs, breast, and scrotum, and can progress to permanent swelling of the legs or arms called elephantiasis. Mp can cause itching, swelling, fever, headache, or other symptoms. Ivermectin and albendazole are medicines used to treat lymphatic filariasis. They eliminate the Wb parasite from the blood but do not affect Mp. Doxycycline is used to treat many kinds of infections and has also recently been shown to reduce the number of filarial worms in several types of filarial infections. The drug may be useful in Mp infections as well.

Residents of Sabougou and nearby villages in Mali who are infected with the Mp parasite, are between 14 and 65 years of age, are in good health, are not pregnant or breastfeeding, and weigh at least 40 kg (88 lb) may be eligible for this study. They may or may not also be infected with Wb. Candidates are screened with a brief medical history and physical examination and blood tests to look for infection with Mp and Wb.

Participants undergo a complete physical examination and medical history. Blood is drawn for routine blood tests. Participants are then randomly assigned to one of four treatment groups, as follows: 1) doxycycline for 6 weeks; 2) doxycycline for 6 weeks followed by a single dose of albendazole and ivermectin given 6 months after the beginning of doxycycline treatment; 3) a single dose of albendazole and ivermectin given 6 months after the beginning of doxycycline treatment; or 4) no treatment. Only patients infected with Wb receive albendazole and ivermectin treatment.

All participants, whether or not they receive doxycycline, come to the clinic every day for 6 weeks. Every 2 weeks during this time, they have a blood test and, in women of childbearing age, a urine pregnancy test. After 6 months, they have a medical history, physical examination, and blood tests. Subjects in the albendazole/ivermectin treatment group are given the pills to take at that time. One year and three years after beginning the study, participants return to the clinic for a final history, physical examination, and blood tests.

At the end of the first year of the study, all participants who tested positive for lymphatic filariasis but did not receive ivermectin and albendazole will be offered treatment with these medicines Ivermectin and albendazole will also be distributed by the Mali government to everyone in the villages as part of a program to eliminate lymphatic filariasis in the country.

DETAILED DESCRIPTION:
Mansonella perstans (Mp) infection is common in areas of Africa that are endemic for Wuchereria bancrofti (Wb), a causative agent of lymphatic filariasis. The clinical and immunologic contributions of Mp infection in this setting are unknown, in part because of the lack of response of Mp to standard antifilarial therapies. The recent discovery of bacterial endosymbionts (Wolbachia) in a number of filarial species, including Mp, has led to new therapeutic options for reducing microfilaremia. Volunteers between the ages of 14 and 65 will be screened in order to identify 240 volunteers (160 Wb+Mp+ and 80 Wb-Mp+) for participation in an open label randomized trial of doxycycline (200 mg daily for 6 weeks). Wb+Mp+ subjects will then be randomized to receive single dose treatment with albendazole and ivermectin 4 months after completion of the doxycycline treatment or no further treatment. Clinical, parasitologic and immunologic assessments will be performed prior to the initiation of treatment and at 6 months and 1 year and 3 years following initiation of treatment. The efficacy of doxycycline treatment in reducing Mp microfilaremia will be assessed in subjects with and without Wb coinfection. In addition, the effect of subsequent administration of albendazole/ivermectin on Mp clearance will be assessed in coinfected subjects.

ELIGIBILITY:
* INCLUSION CRITERIA - SCREENING:

Age 14 to 65.

Both genders.

Not pregnant or breastfeeding by history.

EXCLUSION CRITERIA - SCREENING:

Non-volunteers.

Age less than 14 or greater than 65.

Pregnant or breastfeeding by history.

INCLUSION CRITERIA - TREATMENT:

Age 14 to 65 years.

Men and non-pregnant or breastfeeding women.

EXCLUSION CRITERIA - TREATMENT:

Non-volunteers.

Age less than 14 or greater than 65.

Pregnancy or breast-feeding.

Hgb less than or equal to 10 g/dl.

Cr greater than 1.4/100 ml.

ALT greater than 45 U or bilirubin greater than 1.5.

Weight less than 40 kg.

Heavy alcohol use (more than 1 beer or other alcohol-containing drink/day).

Temperature greater than 37.5C or other serious medical illnesses.

History of allergy to doxycycline or other tetracyclines.

History of HIV infection or other immunocompromised state.

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1500
Dates: Start 2004-12-06; Primary Completion 2007-10-04 (Actual)

PRIMARY OUTCOMES:
Greater than or equal to 50 percent of Mp microfilaremia at 1 year in response to doxycycline treatment in study volunteers with Mp infection.

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Allergy and Infectious Diseases (NIAID), 9000 Rockville Pi, Bethesda, Maryland, United States

REFERENCES:
- [Background] Beach MJ, Streit TG, Addiss DG, Prospere R, Roberts JM, Lammie PJ. Assessment of combined ivermectin and albendazole for treatment of intestinal helminth and Wuchereria bancrofti infections in Haitian schoolchildren. Am J Trop Med Hyg. 1999 Mar;60(3):479-86. doi: 10.4269/ajtmh.1999.60.479. PMID 10466981
- [Background] Addiss DG, Beach MJ, Streit TG, Lutwick S, LeConte FH, Lafontant JG, Hightower AW, Lammie PJ. Randomised placebo-controlled comparison of ivermectin and albendazole alone and in combination for Wuchereria bancrofti microfilaraemia in Haitian children. Lancet. 1997 Aug 16;350(9076):480-4. doi: 10.1016/S0140-6736(97)02231-9. PMID 9274584
- [Background] Horton J, Witt C, Ottesen EA, Lazdins JK, Addiss DG, Awadzi K, Beach MJ, Belizario VY, Dunyo SK, Espinel M, Gyapong JO, Hossain M, Ismail MM, Jayakody RL, Lammie PJ, Makunde W, Richard-Lenoble D, Selve B, Shenoy RK, Simonsen PE, Wamae CN, Weerasooriya MV. An analysis of the safety of the single dose, two drug regimens used in programmes to eliminate lymphatic filariasis. Parasitology. 2000;121 Suppl:S147-60. doi: 10.1017/s0031182000007423. PMID 11386686
- [Derived] Coulibaly YI, Dembele B, Diallo AA, Lipner EM, Doumbia SS, Coulibaly SY, Konate S, Diallo DA, Yalcouye D, Kubofcik J, Doumbo OK, Traore AK, Keita AD, Fay MP, Traore SF, Nutman TB, Klion AD. A randomized trial of doxycycline for Mansonella perstans infection. N Engl J Med. 2009 Oct 8;361(15):1448-58. doi: 10.1056/NEJMoa0900863. PMID 19812401